CLINICAL TRIAL: NCT05985642
Title: An Observational Post-Intervention Control Destination Cohort
Brief Title: Observational PIC Destination Cohort
Status: Recruiting | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5385; UM1AI068636 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-08-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational PIC Destination Cohort: Step 1: Continued analytical treatment interruption (ATI) - During Step 1, PICs will be monitored for safety (including liver function, creatinine, pregnancy, and STI testing), viral, immune, neuropsychological, and socio-behavioral outcomes for up to 96 weeks of continued ATI.
  Step 2: ART Restart - Participants will begin Step 2 if they meet ART restart criteria or reach week 96. Participants will be monitored for safety (including liver function, creatinine, and pregnancy), immune, viral, neuropsychological, and socio-behavioral outcomes through 48 weeks after ART restart.

SUMMARY:
This study is being done to see if people who control HIV without antiretroviral therapy (ART) after receiving an intervention can remain off ART safely. The information collected in this study is also being used to try to understand how people control HIV without ART after receiving an intervention.

DETAILED DESCRIPTION:
This study is a two-step non-interventional study for participants who achieved prolonged viral control off ART, post-intervention (post-intervention control [PIC]) in qualifying AIDS Clinical Trials Group (ACTG) and non-ACTG interventional cure trials (parent studies).

ELIGIBILITY:
Step 1 Inclusion Criteria:

* Currently or previously enrolled in a qualifying ACTG or non- ACTG parent study of curative or suppressive HIV therapy that included an ATI.
* If feasible, participants should not remain co-enrolled in their respective parent study after entering A5385.
* Achieved at least 24 weeks of HIV virus suppression (as defined by the parent study) following ATI initiation, remains off ART with <4 consecutive weeks of HIV-1 RNA >1000 copies/mL, CD4+ T-cell count > 350 cells/mm3 and not experiencing symptoms of acute retroviral syndrome.

NOTE: Participants whose participation has ended on the parent study may still qualify if they have not resumed ART, meet A5385's eligibility criteria, and have not met A5385 ART restart criteria.

* CD4+ T cell count >350 cells/mm3 obtained within 28 days prior to study entry at any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any network-approved non-US laboratory that is IQA certified.
* Willingness to continue ATI for up to 96 weeks or until ART restart criteria are met, and to remain in follow up for 48 weeks after ART restart.
* For participants who are able to become pregnant, negative serum or urine pregnancy test within 24 hours prior to study entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.

NOTE A: Participants who are able to become pregnant are individuals who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, and who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy, tubal ligation, or bilateral salpingectomy.

NOTE B: Acceptable documentation of hysterectomy and bilateral oophorectomy, tubal ligation, and tubal micro-inserts: written documentation or oral communication from a clinician or clinician's staff documented in source documents (physician report/letter, operative report or other source documentation in the patient record, discharge summary, laboratory report, etc.). Participant-reported history is acceptable for documentation of menopause.

* Participants who are able to become pregnant and are engaging in sexual activity that could lead to pregnancy must agree to use one highly effective method of contraception throughout the course of the study from the list below.

Acceptable methods of contraception include:

* Barrier method
* Contraceptive subdermal implant
* Intrauterine device or intrauterine system
* Combined estrogen and progestogen oral contraceptive
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Male partner sterilization with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant.

  * Willingness to use barrier protection (male or female) during sexual activity with all partners not on effective pre-exposure prophylaxis (PrEP) throughout Step 1 ATI and until viral re-suppression in Step 2.

NOTE: Effective PrEP includes ART treatment for partners living with HIV infection.

* Ability and willingness of participant to provide informed consent.

Step 2 Inclusion Criteria:

* Met A5385 ART restart criteria in Step 1.
* Willingness to use barrier protection (male or female) during sexual activity with all partners not on effective PrEP until viral re-suppression.

NOTE: Effective PrEP includes ART treatment for partners living with HIV infection.

Step 1 Exclusion Criteria:

* Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during continued ATI.
* Medical or psychiatric condition (including pregnancy or breastfeeding) that, in the opinion of the site investigator, would place the participant at higher risk of morbidity or would interfere with adherence to study requirements.

NOTE: Site investigators should exercise caution in invoking these criteria and instead aim to support potential participants who are interested and otherwise eligible to participate in the study.

Step 2 Exclusion Criteria:

* Medical or psychiatric condition that, in the opinion of the site investigator, would place the participant at higher risk of morbidity or would interfere with adherence to study requirements.

NOTE: Site investigators should exercise caution in invoking these criteria and instead aim to support potential participants who are interested and otherwise eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who achieved prolonged viral control off ART post-intervention (post-intervention control [PIC]) in qualifying ACTG and non-ACTG interventional cure trials (parent studies).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2029-07-03 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an SAE or Grade ≥3 AE that is related to ATI | From study entry to 96 weeks
  The proportion of participants reporting a serious adverse event (SAE) or a grade ≥ 3 adverse event (AE) that was judged by the A5385 clinical management committee to be at least possibly related to ATI during Step 1.
  An AE is any unfavorable and unintended sign, symptom, or diagnosis occurring in a study participant during the conduct of the study regardless of the attribution. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation or existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or require intervention to prevent one of the outcomes listed above.
  Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Change in CD4 percentage from parent study (pre-ATI) to Step 1 timepoints | From study entry to 96 weeks
  Changes in CD4 percentage (CD4%) are calculated as the CD4% at the specified Step 1 timepoint minus the CD4% measured at the pre-ATI timepoint in the qualifying parent study.
Occurrence of new diagnoses of interest | From study entry through 144 weeks
  Occurrence of new diagnoses of interest during Step 1 and Step 2.
Time from ATI to sustained HIV-1 RNA ≥1000 copies/mL | From study entry to 96 weeks
  Time from ATI to sustained HIV-1 RNA ≥1000 copies/mL over a 4-week period during Step 1.
HIV RNA below 200 copies/mL | 24 weeks after re-starting ART
  The proportion of participants with HIV RNA below 200 copies/mL at 8, 12, and 24 weeks after ART restart.
Change in CD4% from pre-ATI to Step 2 | From study entry to Step 2 week 24
  Change in CD4% from pre-ATI (parent study) to Step 2 Week 12 and Step 2 Week 24 (after ART restart).
Measurements of reservoir | From 24 weeks to 48 weeks after ART restart
  Measurements of reservoir [e.g., intact proviral DNA assay (IPDA)] every 24 weeks during ATI, and 24 and 48 weeks after ART restart.

SECONDARY OUTCOMES:
Time from ATI to ART restart due to a viral, immune, or clinical reason | From study entry to 96 weeks
  Time from ATI to ART restart due to a viral reason (plasma HIV-1 RNA ≥1000 copies/mL for ≥4 consecutive weeks without at least a 0.2 log10 decline from the previous week), and immune reason (confirmed CD4+ T cell count <350), or a clinical reason (e.g., acute retroviral syndrome).
Time from ATI to ART restart | From study entry to 96 weeks
  Time from ATI to ART restart, for any reason.
Measurement of circulating reservoir | Every 24 weeks in Step 1 (up to 96 weeks) and Step 2 Week 24 and 48
  Cell-associated HIV-1 DNA and HIV-1 RNA measured in CD4+ T cells.
Plasma HIV-1 RNA at each study visit | From study entry to 144 weeks
  Plasma HIV-1 RNA (copies/mL) at each study visit measured by clinical assay, or if unquantifiable by standard clinical assay (e.g., below the limit of quantification), single copy assay.
Measurement of replication-competent virus | Every 24 weeks in Step 1 (up to 96 weeks) and Step 2 Week 24 and 48
  Replication-competent virus, measured by the QVOA assay (or appropriate reservoir assay at time of testing).

OTHER OUTCOMES:
Biomarkers of systemic inflammation and immune activation | From 24 weeks to 48 weeks after ART restart
  Measurements of plasma soluble biomarkers of systemic inflammation and immune activation every 24 weeks during ATI and at 24 and 48 weeks after ART restart.
Anti-HIV cellular humoral and innate responses | From 24 weeks to 48 weeks after ART restart
  Anti-HIV cellular humoral and innate responses every 24 weeks during ATI and at 24 and 48 weeks after ART restart.
Association of viral or host characteristics with time to ART restart | From study entry to 96 weeks
  Viral or host characteristics, including, but not limited to, laboratory measures (e.g., viral, inflammatory, reservoir, immune measures), host genetics (e.g., CCR5 heterogeneity, HLA type), or host demographics (e.g., gender, biologic sex, age) for association with time to meeting HIV-1 related, or any, ART restart criteria.
Virus properties and immune responses surrounding time of viral rebound | From study entry to 96 weeks
  Properties of rebound virus, including genotype and phenotype by relevant assays, and immune response surrounding time of viral rebound.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Bar, MD, Study Chair — Penn Therapeutics Clinical Research Site
Locations (4):
- United States (4):
  - University of California, San Francisco HIV/AIDS CRS (801), San Francisco, California
  - Washington University Therapeutics (WT) CRS (2101), St Louis, Missouri
  - Weill Cornell Upton CRS (7803), New York, New York
  - Case CRS (2501), Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Acknowledgement before receiving the data.